CLINICAL TRIAL: NCT02510950
Title: A Pilot Study to Assess the Safety, Feasibility, and Preliminary Efficacy of a Neoepitope-based Personalized Vaccine Approach in Patients With Newly Diagnosed Glioblastoma
Brief Title: Neoepitope-based Personalized Vaccine Approach in Patients With Newly Diagnosed Glioblastoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Low accrual
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201510022
Record Dates: First submitted 2015-07-27; First posted 2015-07-29 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Glioblastoma Multiforme; Astrocytoma, Grade IV
MeSH Terms: conditions — Glioblastoma | interventions — poly ICLC; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm 1: Peptide/poly-ICLC (Experimental): * For all patients, concurrent chemoradiation with temozolomide will be given per standard of care and is outside the scope of this study as per standard of care.
  * The long peptide + poly-ICLC will be given on Cycle 1 Day 1 of maintenance temozolomide.
  * If the vaccine is not ready by this time, the first vaccination will begin on Day 1 of the next cycle of maintenance temozolomide.
  * The peptide + poly-ICLC vaccine will be given again on Days 8, 15, and 22 of the first cycle, as a priming strategy.
  * On all subsequent cycles, the peptide vaccine + poly-ICLC will be given on Day 22 (+/-3 days).
  Interventions: Biological: Personalized peptide vaccine; Drug: Poly-ICLC; Drug: Temozolomide

INTERVENTIONS:
Biological: Personalized peptide vaccine
Drug: Poly-ICLC
  Other Names: Hiltonol
Drug: Temozolomide
  Other Names: Temodar®

SUMMARY:
The early clinical development paradigm for chemotherapeutic agents has significantly influenced the development of therapeutic cancer vaccines. However, there are major differences between these two classes of therapeutics that have important implications for early clinical development. Specifically, the phase 1 concept of dose escalation to find a maximum-tolerated dose does not apply to most therapeutic cancer vaccines. Most therapeutic cancer vaccines are associated with minimal toxicity at a range that is feasible to manufacture or administer, and there is little reason to believe that the maximum-tolerated dose is the most effective dose.

In a recent article from the biostatistics literature, Simon et al. write that "the initial clinical trial of many new vaccines will not be a toxicity or dose-ranging trial but rather will involve administration of a fixed dose of vaccine … in most cases the dose selected will be based on preclinical findings or practical considerations. Using several dose levels in the initial study to find the minimal active dose or to characterize the dose-activity relationship is generally not realistic".

Consistent with these recommendations, the general philosophy of the phase 1 clinical trial is to facilitate a prompt preliminary evaluation of the safety and immunogenicity of the personalized synthetic long peptide vaccine strategy. The proposed clinical trial will test a fixed dose of vaccine. There is considerable experience with the synthetic long peptide vaccine platform. The synthetic long peptide vaccine platform has an excellent safety profile, and the optimal dose appears to be based on practical considerations (solubility of the peptide). The dose to be tested in the proposed clinical trial is consistent with other similar cancer vaccine trials that have been recently completed or are currently ongoing. The sample size (n=10) will provide a reasonably reliable estimate of the safety and immunogenicity of the vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed histologically confirmed glioblastoma multiforme (WHO grade IV). Patients with secondary glioblastoma, in particular those who are IDH1 or IDH2 mutant, will not be excluded.
* Patients who had craniotomy with biopsy, subtotal resection, total gross resection, or re-resection will be permitted.
* Consented to genome sequencing and dbGaP-based data sharing and has provided or will provide germline (PBMC) and tumor DNA/RNA samples of adequate quality for sequencing. (Acquisition of specimens for sequencing and the sequencing itself may be done under this study or as part of routine care or another research project.)
* At least 18 years of age.
* Karnofsky performance status ≥ 60%
* Normal bone marrow and organ function as defined below:

  * Absolute neutrophil count ≥ 1,500/mcL
  * Platelets ≥ 100,000/mcL
  * Total bilirubin ≤ 1.5 x IULN
  * AST(SGOT)/ALT(SGPT) ≤ 3.0 x IULN
  * Creatinine ≤ IULN OR creatinine clearance ≥ 60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
* Systemic corticosteroid therapy is permitted provided dosing is no greater than 4 mg per day (dexamethasone or equivalent) on the day of vaccine administration
* Bevacizumab will be allowed if given for symptomatic control of vasogenic edema and to avoid high dose of corticosteroids
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* As this is a safety and feasibility study, prior immunotherapy will be permitted. However, any prior immunotherapy must be discontinued at least 2 weeks before peptide vaccine administration. Non-immunologic therapy may be continued.
* Inadequate tissue acquisition to allow for neoantigen screening
* No candidate neoantigen identified during screening
* A history of other malignancy ≤ 3 years previous with the exception of non-melanoma skin cancer, any in situ cancer that has been successfully resected and cured, treated superficial bladder cancer, or any early-stage solid tumor that was successfully resected without need for adjuvant radiation or chemotherapy.
* Currently receiving any other investigational agents.
* Known allergy, or history of serious adverse reaction to, vaccines such as anaphylaxis, hives, or respiratory difficulty.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to poly-ICLC or other agents used in the study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* History of pre-existing immunodeficiency disorder including chronic infection (i.e. hepatitis B, hepatitis C, HIV), or autoimmune condition requiring immunosuppressive therapy. This includes inflammatory bowel disease, ulcerative colitis, Crohn's disease, systemic vasculitis, scleroderma, psoriasis, multiple sclerosis, hemolytic anemia, immune-mediated thrombocytopenia, rheumatoid arthritis, systemic lupus erythematosus, Sjogren's syndrome, sarcoidosis, or other rheumatologic disease or any other medical condition or use of medication which might make it difficult for the patient to complete the full course of treatments or to generate an immune response to vaccines.
* Presence of clinically significant increased intracranial pressure (e.g. impending herniation) or hemorrhage, uncontrolled seizures, or requirement for immediate palliative treatment.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 7 days of first dose of vaccine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-12-03 (Actual); Primary Completion 2017-02-14 (Actual); Study Completion 2017-02-14 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of adjuvant personalized neoantigen peptide vaccine with poly-ICLC as measured by grade 3 and 4 adverse events as defined by CTCAE v. 4.03 | 30 days after completion of treatment (approximately 7 months)
Feasibility of the peptide vaccine with poly-ICLC as measured by the ability to identify patient tumor-derived candidate neoantigens and generate a tumor-specific vaccine from time of initial diagnosis to time of proposed administration of the vaccine | Approximately 12-14 weeks

SECONDARY OUTCOMES:
Progression-free survival (PFS) rate | Up to 24 months after last dose of vaccine
  * PFS: duration of time from start of treatment to time of progression or death, whichever occurs first.
  * Progression will be evaluated using the updated response assessment criteria for high-grade gliomas: Response Assessment in Neuro-Oncology (RANO) working group guideline
Overall survival (OS) rate | Up to 24 months after last dose of vaccine
  OS: duration of time from start of treatment to time of death from any cause
Number of neoantigens present in patients with newly diagnosed GBM | After completion of treatment (approximately 6 months)

CONTACTS AND LOCATIONS:
Overall Officials: Gavin Dunn, M.D., Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu